CLINICAL TRIAL: NCT02658149
Title: Psoas Compartment Block Versus Periarticular Local Anesthetic Infiltration for Pain Management for Total Hip Arthroplasty: A Prospective, Randomized Study
Brief Title: Psoas Compartment Block Versus Periarticular Local Anesthetic for Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, James Verner, MD, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-422
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis; Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Ropivacaine; Epinephrine; Morphine; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psoas Compartment Block (Experimental): After exposure anesthetic (Ropivacaine with NaCl) is introduced directly into the iliopsoas muscle, where it then spreads to the lumbar plexus (the nerves responsible for sensation around the surgical site).
  Interventions: Drug: Ropivacaine with NaCl
- Periarticular Local Anesthetic (Active Comparator): An anesthetic "cocktail" of four drugs (ropivacaine, epinephrine, ketorolac tromethamine, morphine) is injected at five locations at the surgical site to the surrounding tissues.
  Interventions: Drug: Epinephrine; Drug: Morphine; Drug: Ketorolac Tromethamine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine with NaCl — 50 mL (40 mL of 0.2% Ropivicaine and 10 mL of 0.9% NaCl) are administered into the psoas compartment
  Other Names: Naropin with NaCl
  Arms: Psoas Compartment Block
Drug: Epinephrine — 0.15 mg Epinephrine are injected as part of the drug "cocktail"
  Other Names: adrenaline
  Arms: Periarticular Local Anesthetic
Drug: Morphine — 4 mg Morphine are injected as part of the drug "cocktail"
  Arms: Periarticular Local Anesthetic
Drug: Ketorolac Tromethamine — 30 mg morphine are injected as part of the drug "cocktail"
  Other Names: Toradol
  Arms: Periarticular Local Anesthetic
Drug: Ropivacaine — 30 mL 0.5% Ropivicaine are injected as part of the drug "cocktail"
  Other Names: Naropin
  Arms: Periarticular Local Anesthetic

SUMMARY:
The primary objective of this study is to examine whether there is a difference in the level of resting pain following total hip arthroplasty with an anterior approach with use of a psoas compartment block versus a local periarticular anesthetic infiltration

DETAILED DESCRIPTION:
A single-center, prospective, randomized clinical trial with a total of 100 patients. One orthopaedic adult reconstruction surgeon at Beaumont Hospital Royal Oak (JJV) will perform all surgeries. After the patient has consented they will be randomized to one of the following two groups:

1. Psoas compartment block (n=50)
2. Periarticular local anesthetic infiltration (n=50),

The patient will be blinded to the study group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary total hip arthroplasty by Dr. James Verner at Beaumont Hospital Royal Oak
* Have a diagnosis of primary osteoarthritis (i.e. degenerative joint disease)
* Surgical approach is anterior

Exclusion Criteria:

* Minors (age less than 18 years)
* Pregnant (surgically sterile, post-menopausal, or negative blood test)
* Previous ipsilateral hip surgery
* Lumbar instrumentation
* Acute trauma
* Rheumatoid arthritis
* Avascular necrosis
* Hip dysplasia
* Known sensitivity, allergy, or contraindication to anesthetics being used in the study
* Narcotic sensitivity
* History of over 6 months of opioid dependency prior to surgery (excluding tramadol)
* Peripheral neuropathy
* Mental/cognitive impairment that would interfere with the patient's self-assessments of function, pain, or quality of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05-11 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Verner, MD, Principal Investigator — William Beaumont Health
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
Started | 50 | 50
Completed | 49 | 50
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8) | 68 (8) | 67 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 23 | 28 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 47 | 46 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 50 | 99
Preoperative Pain Score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Pain Score; 0=no pain, 10=maximum pain
  units on a scale | 3.4 (2.5) | 2.5 (2.6) | 2.9 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 3 Hours
Description: Visual Analog Scale 0-10; 0 = no pain, 10 = worst pain
Time Frame: 3 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
Number analyzed (Participants) | 49 | 50
units on a scale | 4.0 (2.2) | 2.9 (2.2)
Statistical Analysis 1: Comparison: Psoas Compartment Block vs Periarticular Local Anesthetic; Test type: Other; p = 0.036, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Score at 3-24 Hours
Description: Visual Analog Scale 0-10; 0 = no pain, 10 = worst pain
Time Frame: measured once during time frame 3 hours-24 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
Number analyzed (Participants) | 49 | 50
units on a scale | 1.9 (1.7) | 1.3 (1.4)
Statistical Analysis 1: Comparison: Psoas Compartment Block vs Periarticular Local Anesthetic; Test type: Other; p = 0.204, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain Score at 24-48 Hours
Description: Visual Analog Scale 0-10; 0 = no pain, 10 = worst pain
Time Frame: measured once during time froma 24-48 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
Number analyzed (Participants) | 49 | 50
units on a scale | 1.9 (1.7) | 1.7 (1.7)
Statistical Analysis 1: Comparison: Psoas Compartment Block vs Periarticular Local Anesthetic; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Opioid Usage In-hospital at 24 Hours
Description: Total amount of opioids used per patient (measured with Morphine Equivalent Units)
Time Frame: 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Units (Oral)
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
Number analyzed (Participants) | 49 | 50
Morphine Equivalent Units (Oral) | 19.5 (12.8) | 16.7 (13.6)
Statistical Analysis 1: Comparison: Psoas Compartment Block vs Periarticular Local Anesthetic; Test type: Other; p = 0.741, t-test, 2 sided

5. Secondary Outcome: Opioid Usage In-hospital at 48 Hours
Description: Total amount of opioids used per patient (measured with Morphine Equivalent Units)
Time Frame: 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: Morphine Equivalent Units (Oral)
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
Number analyzed (Participants) | 49 | 50
Morphine Equivalent Units (Oral) | 22.3 (16.8) | 20.8 (16.4)
Statistical Analysis 1: Comparison: Psoas Compartment Block vs Periarticular Local Anesthetic; Test type: Other; p = 1.0, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Psoas Compartment Block | Periarticular Local Anesthetic
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 5/49 | 1/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psoas Compartment Block (N=49) | Periarticular Local Anesthetic (N=50)
Prolonged transient numbness (Nervous system disorders) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study include single surgeon and single institution data, which affects generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT02658149/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02658149/Prot_SAP_001.pdf